CLINICAL TRIAL: NCT04134897
Title: A Multicenter Prospective Phase III Clinical Trial of Neoadjuvant CapOx in Patients With Intermediate Risk CRM-negative Middle Rectal Cancer
Brief Title: Neoadjuvant Chemotherapy in Patients With Moderate Risk Mid Rectal Cancer
Acronym: RuCorT-02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Sergey Gordeyev, Principal Investigator, Consultant surgeon, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RuCorT-02
Record Dates: First submitted 2019-10-19; First posted 2019-10-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Rectal Neoplasms Malignant; Rectum Carcinoma; Rectal Cancer
Keywords: rectal cancer; neoadjuvant chemotherapy; neoadjuvant radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy (Experimental): Patients will receive 4 cycles of neoadjuvant CapOx chemotherapy (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 bid per os days 1-14 every 3 weeks). In case of partial response or stable disease (based on pelvic MRI) patients proceed to surgery within 2 weeks. In case of disease progression patients receive 50 Gy pelvic chemoradiotherapy with capecitabine 825 mg/m2 bid per os on radiation days and then surgery following 8-10 weeks. After surgery patients receive 4 cycles of adjuvant CapOx chemotherapy (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 bid per os days 1-14 every 3 weeks).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy; Procedure: Rectal cancer surgery
- Neoadjuvant radiotherapy (Active Comparator): Patients will receive 5x5 Gy radiotherapy and then surgery following 6-8 weeks. After surgery patients receive 8 cycles of adjuvant CapOx chemotherapy (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 bid per os days 1-14 every 3 weeks).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Procedure: Rectal cancer surgery; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine — 2000 mg/m2, bid, per os, days 1-14, 4 cycles
  Other Names: Xeloda
Drug: Oxaliplatin — 130 mg/m2 iv day 1, 4 cycles
Drug: Capecitabine — 825 mg/m2, bid, per os, only on days of radiation (Monday through Friday)
  Other Names: Xeloda
  Arms: Neoadjuvant chemotherapy
Radiation: Radiotherapy — Pelvic radiotherapy dose: 44 Gy on regional nodes, 50 Gy on primary tumor
  Arms: Neoadjuvant chemotherapy
Procedure: Rectal cancer surgery — Laparoscopic or open total mesorectal excision
Radiation: Radiotherapy — Pelvic radiotherapy dose: 25 Gy in 5 Gy fractions
  Arms: Neoadjuvant radiotherapy

SUMMARY:
The purpose of this study is to determine whether 3 months of neoadjuvant CapOx is non-inferior to neoadjuvant radiotherapy in patients with moderate risk CRM"-" mid rectal cancer.

DETAILED DESCRIPTION:
This trial aims to investigate the efficacy of neoadjuvant chemotherapy compared to 5x5 Gy neoadjuvant radiotherapy in moderate risk CRM-negative rectal cancer patients. This is a prospective multicenter open-label non-inferiority randomized phase III clinical trial. Patients will be randomized using an online randomization system to receive either 4 cycles of neoadjuvant CapOx (oxaliplatin 130 mg/m2 iv day 1, capecitabine 2000 mg/m2 per os bid days 1-14) chemotherapy, surgery and 4 cycles of adjuvant CapOx chemotherapy or 5x5 Gy radiotherapy, surgery and 8 cycles of adjuvant CapOx chemotherapy. A stratification will be performed based on сN stage and clinical center. Patients with сT3c-T3dN0-1M0, cT1-T3dN2M0 cancer in the middle rectum are included. Chemoradiotherapy (50 Gy with concomitant capecitabine 825 mg/m2 per os bid on radiation days) will be performed for patients with tumor progression after neoadjuvant chemotherapy. The main hypothesis is that the 2-year local recurrence rate is non-inferior after neoadjuvant chemotherapy and neoadjuvant radiotherapy in moderate risk mid rectal cancer patients. The target accrual is 158 patients in each treatment arm (including 10% potential data loss) based on non-recurrence rate of 98% in investigated and 96% in the control group with a non-inferiority margin of 3%, α=0,05, power 80%. An interim analysis is planned after 50% of the patients will reach a 2-year followup. Pelvic Magnetic Resonance Imaging (MRI) is performed in all patients for staging before and after neoadjuvant chemotherapy and before surgery. Pelvic MRI is subject to central review. Conduction of this study and data collection are controlled by a local institutional board.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically verified colon rectal adenocarcinoma
* сT3c-T3dN0-1M0, cT1-T3dN2M0. cancer of the middle rectum (based on pelvic MRI)
* Tumor more than 2 mm from mesorectal fascia (based on pelvic MRI)
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* Haemoglobin (HGB) > 90 g/L
* Platelet Count (PLT) > 120x10*9/L
* Serum creatinine < 150 µmol/L
* Total bilirubin < 25 µmol/L

Exclusion Criteria:

* inability to obtain informed consent
* distant metastases
* synchronous or metachronous tumors
* previous chemotherapy or radiotherapy
* clinically significant cardiovascular disorders (myocardial infarction < 6 months before visit, stroke < < 6 months before visit, instable angina < 3 months before visit, arrhythmia, uncontrolled hypertension > 160/100 mm hg
* clinically significant neurological disorders
* previous neuropathy 2 or higher
* current infection or heavy systemic disease
* pregnancy, breastfeeding
* ulcerative colitis
* individual intolerance to treatment components
* proven dihydropyrimidine dehydrogenase (DPD) deficiency
* participation in other clinical trials
* psychiatric disorders, which render patient unable to follow instructions or understand his/her condition
* technical inability to perform pelvic MRI
* inability of long-term followup of the patient
* HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
2-year local recurrence rate | 2 years

SECONDARY OUTCOMES:
Adjuvant chemotherapy compliance | 6 months
  Proportion of patients who receive a complete course of adjuvant chemotherapy
Acute chemotherapy toxicity | 6 months
  Toxicity measured according to NCI-CTCAE v.5.0
pathologic complete response rate (pCR) | 1 month
2-year overall survival | 2 years
2-year disease-free survival | 2 years
Operative morbidity | 30 days
  Morbidity measured according to Clavien-Dindo classification
Neoadjuvant chemotherapy disease progression rate | 3 months
  Proportion of patients with disease progression during neoadjuvant chemotherapy
Preoperative tumor-associated complications rate | 3 months
  The rate of tumor-associated complications (bowel obastruction, bleeding etc) during neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Zaman Z Mamedli, PhD, Principal Investigator — N.N.Blokhin Russian Cancer Research Center
Locations (1):
- N.N.Blokhin Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No